CLINICAL TRIAL: NCT00908310
Title: A Post-marketing Safety Study in Patients With Moderate Renal Insufficiency Who Receive OMNISCAN (Gadodiamide Injection) for Contrast-enhanced Magnetic Resonance Imaging.
Brief Title: Post-marketing Safety Study in Patients With Moderate Renal Insufficiency Who Receive Omniscan for Contrast-enhanced Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GE-041-075
Record Dates: First submitted 2009-05-13; First posted 2009-05-25 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease; Renal Insufficiency
Keywords: CKD - Chronic Kidney Disease; GBCA - Gadolinium-based contrast agent; GFR - Glomerular Filtration Rate; MRI - Magnetic Resonance Imaging; NSF - Nephrogenic Systemic Fibrosis; Known or suspected CKD with an eGFR greater than or equal to 30mL & less than 60 mL/min/1.73m2 as measured within 30 days prior to the OMNISCAN.
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — gadodiamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omniscan (Other)
  Interventions: Drug: Omniscan

INTERVENTIONS:
Drug: Omniscan — OMNISCAN will be administered intravenously at the medical discretion of the prescribing physician.
  Other Names: Gadodiamide

SUMMARY:
This will be an international, multi-center, post-marketing surveillance study in patients with moderate renal insufficiency who are administered gadodiamide, Omniscan, during a MRI. Omniscan will be administered intravenously at the medical discretion of the prescribing physician.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been referred for a clinically indicated MRI examination with a gadolinium-based contrast agent.
* The subject has known or suspected chronic kidney disease with an eGFR greater than or equal to 30mL and <60 mL/min/1.73 m2 as measured within 30 days prior to the planned index OMNISCAN administration.
* The subject agrees to be contacted for follow-up for 24 months.

Exclusion Criteria:

* Patients with known or suspected NSF based on biopsy confirmation or the onset of signs and symptoms of NSF lasting at least 7 days as follows:

  1. skin - swelling, hardening and tightening; reddened or darkened patches; burning or itching;
  2. eyes - yellow raised spots on whites of eyes; or
  3. bones and muscle - stiffness in joints; difficulty in moving or straightening of arms, hands, legs or feet; bone pain especially in hips and ribs or muscle weakness.
* Patients allergic to any GBCA.
* Patients with chronic renal disease with a GFR <30 mL/min/1.73 m2 as measured within 30 days prior to the planned OMNISCAN administration.
* Patients with acute renal insufficiency of any severity due to the hepato-renal syndrome or in the peri operative liver transplantation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, MD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 213 subjects enrolled in this study. Total of 202 subjects evaluated for safety purposes. Total of 153 subjects completed this study. Total of 11 subjects discontinued prior to contrast administration (no contrast media received).
Groups:
- Omniscan: OMNISCAN 287mg/mL will be administered intravenously at the medical discretion of the prescribing physician.
Period: Overall Study
Arm/Group | Omniscan
Started | 213
Completed | 153
Not Completed | 60
Not completed — Death | 37
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 7
Not completed — Screening failure | 5
Not completed — Other reasons | 4

BASELINE CHARACTERISTICS:
Population: The 202 subjects that received contrast media were evaluated for safety.
Arm/Group | Omniscan
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (12.41)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 126
Region of Enrollment [Number; unit: participants]
  United States | 13
  Canada | 28
  China | 62
  India | 10
  Spain | 12
  Taiwan | 77

OUTCOME MEASURES:

1. Primary Outcome: Capture of Post-marketing Safety Information in Patients With Moderate Renal Insufficiency Undergoing Routine Contrast-enhanced MRI With Administration of OMNISCAN in Order to Assess the Risk for Developing Nephrogenic Systemic Fibrosis (NSF).
Description: Capture of safety information in moderate renal insufficiency patients undergoing routine contrast-enhanced MRI with administration of OMNISCAN.
Time Frame: Greater than or equal to 7 days post contrast administration.
Population: Incidence of Nephrogenic Systemic Fibrosis (NSF)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Omniscan
Number analyzed (Participants) | 202
percentage of subjects
  Reporting of NSF and Symptoms | 3.96 [1.73 to 7.65]
  Diagnosis of NSF | 0.00 [0.00 to 1.81]
  Biopsy confirmed NSF | 0.00 [0.00 to 1.81]

ADVERSE EVENTS:
Arm/Group | Omniscan
Serious Adverse Events (participants affected / at risk) | 7/202
Other Adverse Events (participants affected / at risk) | 0/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omniscan (N=202)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pterygium (Eye disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As a result of the FDA reference ID: #2954949, subject enrolment was terminated at 213 subjects. All subjects (202 subjects) who received any dose of Omniscan were followed as per protocol until study completion, withdrawal, or lost-to-follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No